CLINICAL TRIAL: NCT07220018
Title: mHealth Navigation Using SMS Texting to Improve CRC Screening Among Homeless Persons
Brief Title: Colorectal Cancer Screening in the Homeless
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Ramin Asgary, Professor, George Washington University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NCR235230; R01MD019112 (NIH)
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
Keywords: homeless persons; mHealth; short message service; texting
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial evaluating an intervention against a control
Who Masked: Investigator
Masking Description: Data analyst
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colorectal Cancer Specific Education (Experimental): 6 months of mHealth Colorectal cancer educational messages. The content will address elements such as activating and educating patients, exploring and removing challenges, accommodating personal goals, and engaging and targeting subgroups. Texts will be delivered to encourage cancer screenings and lifestyle changes, and participants will receive appointment reminders before each appointment with a follow-up text and robocall if the appointment is missed.
  Interventions: Behavioral: mHealth for Colorectal cancer screening in Homeless Persons
- General Health Education (Other): 6 months of mHealth, including basic healthcare and general health promotion via SMS texts that do not overlap with CRC screening content.
  Interventions: Other: Control SMS Messages

INTERVENTIONS:
Behavioral: mHealth for Colorectal cancer screening in Homeless Persons — Specific colorectal cancer educational SMS text messages are sent to participants' mobile phones
  Arms: Colorectal Cancer Specific Education
Other: Control SMS Messages — Standard health information SMS text messages sent to participants' mobile phones
  Arms: General Health Education

SUMMARY:
This study is designed to assess the effect of implementing a text messaging strategy for colorectal cancer screening among homeless persons aged 45-75 years, who are not up to date on colorectal cancer screening, in shelter clinics in NYC. This mixed-methods study uses a randomized clinical trial design and semi-structured interviews.

DETAILED DESCRIPTION:
This study seeks to evaluate the extent to which an SMS text-based patient navigation will mitigate some of the barriers to and improve CRC screening in homeless persons. It will include processes customized to the homeless specific needs via a streamlined approach of an SMS text-based navigation in shelters clinics to explain cancer risks and screening options, provide test instructions and support, identify and resolve challenges to screening, respond to questions and concerns, make appointments for screening, support screening completion, provide post-screen counselling, and obtain test results to complete screening loop. The target population will be homeless persons aged 45-75, not up-to-date with CRC screening, recruited from shelter clinics of a community organization serving homeless persons in New York City (NYC). The specific aims of this mixed methods study are:

AIM 1: To evaluate the effect of 6-month SMS text-based patient navigation for CRC screening (INT) versus an attention control (CL) of general health promotion on the completion rates of CRC screening using a randomized trial design in shelter clinics. Hypothesis 1) among homeless persons aged 45-75 not up-to-date with CRC screening, those randomized to the INT (n=294) will have higher CRC screening rates in the magnitude of 10 percentage points, compared to those randomized to the CL (n=294) at 6 months post enrollment. Individual-level randomization will be employed in shelter clinics in NYC.

AIM 2: To evaluate perceptions, attitudes, and experiences of homeless persons (n=50) and providers and staff (n=20) on SMS text navigation for CRC screening in shelter clinics using semi-structured interviews. The results will strengthen the SMS navigation approach by revealing barriers and necessary adaptation needs.

AIM 3: To evaluate perceptions and attitudes of program staff (n=20) of agencies servicing homeless persons in NYC and on the national level on challenges and opportunities of implementing SMS text navigation for cancer care and control in the shelter system using semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* Homeless persons aged 45 - 75 years old, with no up-to-date colorectal cancer screening defined as: 1) no colonoscopy in the past 10 years, or 2) no Flexible sigmoidoscopy, Digital Contrast Barium Enema, or CT colonoscopy in the past 5 years, or 3) no Fecal Immunochemical Test/Fecal Occult Blood in the past 12 months or mt-sDNA/Cologuard Test in the past three years
* English or Spanish speaking
* currently presenting to the shelter clinics for medical care
* connected to multidisciplinary social and health services in NYC shelter clinics

Exclusion Criteria:

* known active/uncontrolled illness rendering homeless persons to undergo screening, CRC in the past 2 years, colectomy, Inflammatory Bowel Dis., Familial Adenomatous Polyposis or other colorectal diseases in which screening is different from average CRC risk and methods, inability to consent, serious/significant comorbidity where life expectancy is limited or screening is not recommended, which will be verified by their respective provider
* inability to read and respond to SMS texts
* any condition preventing participants from providing informed consent.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
Completion of CRC Screening | 6 months
  Completed rates of CRC screenings (colonoscopy or FIT test)

SECONDARY OUTCOMES:
Perceptions, Attitudes, and Experiences on SMS texts | 6 months
  Semi-structured Interviews with participants and providers

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Asgary, MD, MPH, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asgary R, Garland V, Jakubowski A, Sckell B. Colorectal cancer screening among the homeless population of New York City shelter-based clinics. Am J Public Health. 2014 Jul;104(7):1307-13. doi: 10.2105/AJPH.2013.301792. Epub 2014 May 15. PMID 24832144
- [Background] Asgary R, Sckell B, Alcabes A, Naderi R, Ogedegbe G. Perspectives of cancer and cancer screening among homeless adults of New York City shelter-based clinics: a qualitative approach. Cancer Causes Control. 2015 Oct;26(10):1429-38. doi: 10.1007/s10552-015-0634-0. Epub 2015 Jul 25. PMID 26208591
- [Background] Asgary R, Sckell B, Alcabes A, Naderi R, Adongo P, Ogedegbe G. Perceptions, Attitudes, and Experience Regarding mHealth Among Homeless Persons in New York City Shelters. J Health Commun. 2015;20(12):1473-80. doi: 10.1080/10810730.2015.1033117. Epub 2015 Aug 27. PMID 26313765
- [Background] Asgary R. Cancer screening in the homeless population. Lancet Oncol. 2018 Jul;19(7):e344-e350. doi: 10.1016/S1470-2045(18)30200-6. Epub 2018 Jun 29. PMID 30084381